CLINICAL TRIAL: NCT05956002
Title: A PHASE 1, OPEN-LABEL, RANDOMIZED, SINGLE DOSE, CROSSOVER STUDY TO ESTIMATE THE RELATIVE BIOAVAILABILITY OF ETRASIMOD (PF-07915503) MINI TABLETS IN WATER AND 3 FOOD VEHICLES COMPARED TO THE ETRASIMOD (PF-07915503) CLINICAL IR TABLETS UNDER FASTED CONDITIONS, AND TO EVALUATE MINI TABLET PALATABILITY IN HEALTHY ADULT PARTICIPANTS
Brief Title: A Study to Evaluate the Study Medication (Etrasimod) When Mixed With Food in Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: C5041034; 2023-504411-32-00 (Registry Identifier: CTIS (EU))
Record Dates: First submitted 2023-06-29; First posted 2023-07-21 (Actual); Results first posted 2025-02-10 (Actual); Last update posted 2025-02-10 (Actual); Status verified 2025-02

CONDITIONS: Healthy Participants
Keywords: bioavailability; etrasimod; adult

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Sequence 1 (Experimental): Single oral dose of etrasimod 2 mg clinical IR tablet under fasted conditions (Reference) followed by single oral dose of etrasimod 2 mg mini tablets mixed with applesauce under fasted conditions (Test 1) followed by single oral dose of etrasimod 2 mg mini tablets mixed with chocolate pudding under fasted conditions (Test 2) followed by single oral dose of etrasimod 2 mg mini tablets mixed with water under fasted conditions (Test 3) followed by single oral dose of etrasimod 2 mg mini tablets mixed with yogurt under fasted conditions (Test 4)
  Interventions: Drug: Estraimod Immediate Release (IR); Drug: Etrasimod Mini Tab in water; Drug: Etrasimod Mini Tab in chocolate pudding; Drug: Etrasimod Mini Tab in yogurt; Drug: Etrasimod Mini Tab in applesauce
- Sequence 2 (Experimental): Single oral dose of etrasimod 2 mg mini tablets mixed with applesauce under fasted conditions (Test 1) followed by single oral dose of etrasimod 2 mg mini tablets mixed with water under fasted conditions (Test 3) followed by single oral dose of etrasimod 2 mg clinical IR tablet under fasted conditions (Reference) followed by single oral dose of etrasimod 2 mg mini tablets mixed with chocolate pudding under fasted conditions (Test 2) followed by single oral dose of etrasimod 2 mg mini tablets mixed with yogurt under fasted conditions (Test 4)
  Interventions: Drug: Estraimod Immediate Release (IR); Drug: Etrasimod Mini Tab in water; Drug: Etrasimod Mini Tab in chocolate pudding; Drug: Etrasimod Mini Tab in yogurt; Drug: Etrasimod Mini Tab in applesauce
- Sequence 3 (Experimental): Single oral dose of etrasimod 2 mg mini tablets mixed with chocolate pudding under fasted conditions (Test 2). Followed by single oral dose of etrasimod 2 mg clinical IR tablet under fasted conditions (Reference).followed by single oral dose of etrasimod 2 mg mini tablets mixed with water under fasted conditions (Test 3). Followed by single oral dose of etrasimod 2 mg mini tablets mixed with applesauce under fasted conditions (Test 1) Followed by single oral dose of etrasimod 2 mg mini tablets mixed with yogurt under fasted conditions (Test 4)
  Interventions: Drug: Estraimod Immediate Release (IR); Drug: Etrasimod Mini Tab in water; Drug: Etrasimod Mini Tab in chocolate pudding; Drug: Etrasimod Mini Tab in yogurt; Drug: Etrasimod Mini Tab in applesauce
- Sequence 4 (Experimental): Single oral dose of etrasimod 2 mg mini tablets mixed with water under fasted conditions (Test 3). Followed by single oral dose of etrasimod 2 mg mini tablets mixed with chocolate pudding under fasted conditions (Test 2). Followed by single oral dose of etrasimod 2 mg mini tablets mixed with applesauce under fasted conditions (Test 1). Followed by single oral dose of etrasimod 2 mg clinical IR tablet under fasted conditions (Reference). Followed by single oral dose of etrasimod 2 mg mini tablets mixed with yogurt under fasted conditions (Test 4)
  Interventions: Drug: Estraimod Immediate Release (IR); Drug: Etrasimod Mini Tab in water; Drug: Etrasimod Mini Tab in chocolate pudding; Drug: Etrasimod Mini Tab in yogurt; Drug: Etrasimod Mini Tab in applesauce

INTERVENTIONS:
Drug: Estraimod Immediate Release (IR) — an immediate release tablet
Drug: Etrasimod Mini Tab in water — very small tablet mixed in water
Drug: Etrasimod Mini Tab in chocolate pudding — very small tablet mixed in chocolate pudding
Drug: Etrasimod Mini Tab in yogurt — Very small tablet mixed in yogurt
Drug: Etrasimod Mini Tab in applesauce — Very small tablet mixed in applesauce

SUMMARY:
The purpose of this study is to compare how healthy adults process Etrasimod when taken in different forms. One form is Etrasimod taken without food. The other form is Etrasimod mixed with water and 3 different foods. The types of food used are applesauce, chocolate pudding or yogurt.

The study is seeking participants who are:

* Aged 18 or older
* Male or female who are healthy as determined by medical assessment
* Body-mass index (BMI) of 16 to 32, and a total body weight > 50kg.

The study will take up to 2.5 months, including the screening period. Participants will have to stay at the study clinic for at least 45 days. This includes 5 study periods in total.

Participants will take Etrasimod as a tablet by mouth without food. Participants will also take Etrasimod sprinkled in soft food or water. Blood samples will be taken both before and after participants take Etrasimod. Participants will also answer questions for taste assessment purposes. A follow-up phone call will be made 20 to 27 days after the last study period.

ELIGIBILITY:
Inclusion Criteria:

* Healthy participants
* BMI 16 to 32 kg/m2
* body weight more than 50kg

Exclusion Criteria:

* Ongoing or past history of significant medical conditions
* Eye disorders such as macular edema or uveitis
* Ongoing or recent infections
* Use of prescription or non prescription medications within 7 days of first dose
* Smoking or using nicotine products equivalent to more than 5 cigarettes per day
* History of severe allergic or anaphylactic reactions

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2023-09-04 (Actual); Primary Completion 2024-01-04 (Actual); Study Completion 2024-01-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer Clinical Research Unit - Brussels, Brussels, Bruxelles-capitale, Région de, Belgium

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=C5041034

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 16 participants were enrolled in this study.
Pre-assignment Details: All participants received at least one dose of etrasimod prepared in different vehicles.
Groups:
- Treatment Sequence: A Then B Then C Then D Then E: Participants were randomized to receive a single oral dose of etrasimod 2 milligram (mg) clinical immediate release (IR) tablet with 240 milliliter (ml) of water on Day 1 of Period 1 under fasted conditions as reference (Treatment A) followed by single oral dose of etrasimod 2 mg mini tablets mixed with 5 ml applesauce (Treatment B) as test 1 on Day 1 of Period 2 followed by single oral dose of etrasimod 2 mg mini tablets mixed with 5 ml chocolate pudding (Treatment C) as test 2 on Day 1 of Period 3 followed by single oral dose of etrasimod 2 mg mini tablets mixed with 5 ml water (Treatment D) as test 3 on Day 1 of Period 4 followed by single oral dose of etrasimod 2 mg mini tablets mixed with 5 ml yogurt (Treatment E) as test 4 on Day 1 of Period 5. There was a washout period of 9 days between each dose.
- Treatment Sequence: B Then D Then A Then C Then E: Participants were randomized to receive a single oral dose of etrasimod 2 mg mini tablets mixed with 5 ml applesauce (Treatment B) as test 1 on Day 1 of Period 2 followed by single oral dose of etrasimod 2 mg mini tablets mixed with 5ml water (Treatment D) as test 3 on Day 1 of Period 4 followed by single oral dose of etrasimod 2 mg clinical IR tablet (Treatment A) as reference with 240 ml of water on Day 1 Period 1 under fasted conditions, followed by single oral dose of etrasimod 2 mg mini tablets mixed with 5ml chocolate pudding (Treatment C) as test 2 on Day 1 of Period 3 followed by single oral dose of etrasimod 2 mg mini tablets mixed with 5 ml yogurt (Treatment E) as test 4 on Day 1 of Period 5. There was a washout period of 9 days between each dose.
- Treatment Sequence: C Then A Then D Then B Then E: Participants were randomized to receive a single oral dose of etrasimod 2 mg mini tablets mixed with 5 ml chocolate pudding (Treatment C) as test 2 on Day 1 of Period 3. Followed by single oral dose of etrasimod 2 mg clinical IR tablet (Treatment A) as reference with 240 ml of water on Day 1 of Period 1 under fasted conditions, followed by single oral dose of etrasimod 2 mg mini tablets mixed with 5 ml water (Treatment D) as test 3 on Day 1 of Period 4 , Followed by single oral dose of etrasimod 2 mg mini tablets mixed with 5 ml applesauce (Treatment B) as test 1 on Day 1 of Period 2, followed by single oral dose of etrasimod 2 mg mini tablets mixed with 5 ml yogurt (Treatment E) as test 4 on Day 1 of Period 5. There was a washout period of 9 days between each dose.
- Treatment Sequence: D Then C Then B Then A Then E: Participants were randomized to receive a single oral dose of etrasimod 2 mg mini tablets mixed with 5 ml water (Treatment D) as test 3 on Day 1 of Period 4. Followed by single oral dose of etrasimod 2 mg mini tablets mixed with 5 ml chocolate pudding (Treatment C) as test 2 on Day 1 of Period 3. Followed by single oral dose of etrasimod 2 mg mini tablets mixed with 5 ml applesauce (Treatment B) as test 1 on Day 1 of Period 2, followed by single oral dose of etrasimod 2 mg clinical IR tablet with 240 ml of water on Day 1 of Period 1 of each period under fasted conditions (Treatment A) as reference. Followed by single oral dose of etrasimod 2 mg mini tablets mixed with 5 ml yogurt (Treatment E) as test 4 on Day 1 of Period 5. There was a washout period of 9 days between each dose.
Period: Treatment Period 1
Arm/Group | Treatment Sequence: A Then B Then C Then D Then E | Treatment Sequence: B Then D Then A Then C Then E | Treatment Sequence: C Then A Then D Then B Then E | Treatment Sequence: D Then C Then B Then A Then E
Started | 4 | 4 | 4 | 4
Completed | 4 | 4 | 4 | 4
Not Completed | 0 | 0 | 0 | 0
Period: Washout Period
Arm/Group | Treatment Sequence: A Then B Then C Then D Then E | Treatment Sequence: B Then D Then A Then C Then E | Treatment Sequence: C Then A Then D Then B Then E | Treatment Sequence: D Then C Then B Then A Then E
Started | 4 | 4 | 4 | 4
Completed | 4 | 4 | 4 | 4
Not Completed | 0 | 0 | 0 | 0
Period: Treatment Period 2
Arm/Group | Treatment Sequence: A Then B Then C Then D Then E | Treatment Sequence: B Then D Then A Then C Then E | Treatment Sequence: C Then A Then D Then B Then E | Treatment Sequence: D Then C Then B Then A Then E
Started | 4 | 4 | 4 | 4
Completed | 4 | 4 | 4 | 4
Not Completed | 0 | 0 | 0 | 0
Period: Washout Period
Arm/Group | Treatment Sequence: A Then B Then C Then D Then E | Treatment Sequence: B Then D Then A Then C Then E | Treatment Sequence: C Then A Then D Then B Then E | Treatment Sequence: D Then C Then B Then A Then E
Started | 4 | 4 | 4 | 4
Completed | 4 | 4 | 4 | 4
Not Completed | 0 | 0 | 0 | 0
Period: Treatment Period 3
Arm/Group | Treatment Sequence: A Then B Then C Then D Then E | Treatment Sequence: B Then D Then A Then C Then E | Treatment Sequence: C Then A Then D Then B Then E | Treatment Sequence: D Then C Then B Then A Then E
Started | 4 | 4 | 4 | 4
Completed | 4 | 4 | 3 | 4
Not Completed | 0 | 0 | 1 | 0
Not completed — Adverse Event | 0 | 0 | 1 | 0
Period: Washout Period
Arm/Group | Treatment Sequence: A Then B Then C Then D Then E | Treatment Sequence: B Then D Then A Then C Then E | Treatment Sequence: C Then A Then D Then B Then E | Treatment Sequence: D Then C Then B Then A Then E
Started | 4 | 4 | 3 | 4
Completed | 4 | 4 | 3 | 4
Not Completed | 0 | 0 | 0 | 0
Period: Treatment Period 4
Arm/Group | Treatment Sequence: A Then B Then C Then D Then E | Treatment Sequence: B Then D Then A Then C Then E | Treatment Sequence: C Then A Then D Then B Then E | Treatment Sequence: D Then C Then B Then A Then E
Started | 4 | 4 | 3 | 4
Completed | 4 | 4 | 3 | 4
Not Completed | 0 | 0 | 0 | 0
Period: Washout Period
Arm/Group | Treatment Sequence: A Then B Then C Then D Then E | Treatment Sequence: B Then D Then A Then C Then E | Treatment Sequence: C Then A Then D Then B Then E | Treatment Sequence: D Then C Then B Then A Then E
Started | 4 | 4 | 3 | 4
Completed | 4 | 4 | 3 | 4
Not Completed | 0 | 0 | 0 | 0
Period: Treatment Period 5
Arm/Group | Treatment Sequence: A Then B Then C Then D Then E | Treatment Sequence: B Then D Then A Then C Then E | Treatment Sequence: C Then A Then D Then B Then E | Treatment Sequence: D Then C Then B Then A Then E
Started | 4 | 4 | 4 (1 participant who temporarily discontinued from study intervention resumed treatment) | 4
Completed | 4 | 4 | 4 | 4
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Safety analysis set (SAS) included all participants who took at least 1 dose of study intervention. Participants were analyzed according to the product they actually received.
Groups:
- All Participants: All participants who were randomized to receive any of the treatment sequence in any of the period were included.
Arm/Group | All Participants
Number analyzed (Participants) | 16
Age, Continuous [Mean (Standard Deviation); unit: Years] | 42.1 (11.27)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 11
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 15
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 11
  More than one race | 0
  Unknown or Not Reported | 2

OUTCOME MEASURES:

1. Primary Outcome: Area Under the Plasma Concentration-Time Curve From Time Zero to the Time of the Last Quantifiable Concentration (AUClast) of Etrasimod
Description: AUClast was calculated using linear/log trapezoidal method.
Time Frame: At pre-dose and 1, 2, 4, 6, 8, 12, 24, 48, 72, 96, 120, 144, and 168 hours post-dose on Day 1 of each period
Population: Pharmacokinetic (PK) parameter analysis set included all participants who took at least 1 dose of study intervention and in whom at least 1 of the PK parameters of interest were reported.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Nanogram*hour per milliliter (ng*hr/mL)
Groups:
- Etrasimod 2 mg IR Tablet: Participants received etrasimod 2 mg IR tablet with volume of 240 ml of water on Day 1 of Period 1, 2, 3 or 4 under fasted conditions.
- Etrasimod 2 mg Mini Tablets in Applesauce: Participants received etrasimod 2mg mini tablets with 5 ml applesauce, followed by approximately 235 mL water on Day 1 of Period 1, 2, 3 or 4 under fasted condition.
- Etrasimod 2 mg Mini Tablets in Chocolate Pudding: Participants received etrasimod 2mg mini tablets with 5 ml chocolate pudding, followed by approximately 235 mL water on Day 1 of period 1, 2, 3 or 4 under fasted condition.
- Etrasimod 2 mg Mini Tablets in Water: Participants received etrasimod 2mg mini tablets with 5 ml water, followed by approximately 235 mL water on Day 1 of Period 1, 2, 3 or 4 under fasted condition.
- Etrasimod 2 mg Mini Tablets in Yogurt: Participants received etrasimod 2mg mini tablets with 5 ml yogurt, followed by approximately 235 mL of water on Day 1 of Period 5 under fasted condition.
Arm/Group | Etrasimod 2 mg IR Tablet | Etrasimod 2 mg Mini Tablets in Applesauce | Etrasimod 2 mg Mini Tablets in Chocolate Pudding | Etrasimod 2 mg Mini Tablets in Water | Etrasimod 2 mg Mini Tablets in Yogurt
Number analyzed (Participants) | 16 | 15 | 16 | 16 | 16
Nanogram*hour per milliliter (ng*hr/mL) | 1620 (26) | 1529 (19) | 1538 (19) | 1391 (22) | 1510 (22)
Statistical Analysis 1: Comparison: Etrasimod 2 mg IR Tablet vs Etrasimod 2 mg Mini Tablets in Applesauce; Analysis was performed for etrasimod 2mg mini tablets in applesauce vs etrasimod 2mg clinical IR tablet mixed effect model with sequence, period and treatment as fixed effects and participant within the sequence as a random effect; Test type: Equivalence — For bioequivalence, the 90% CIs of the adjusted geometric mean ratio of AUClast for etrasimod 2 mg mini tablets mixed with applesauce (tests) compared with etrasimod 2 mg clinical IR tablet (reference) were required to be within the 80 to 125% range; Ratio of adjusted geometric means = 94.66, 90% CI 2-sided [91.33 to 98.12] — The ratio and 90% CIs are expressed as percentages
Statistical Analysis 2: Comparison: Etrasimod 2 mg IR Tablet vs Etrasimod 2 mg Mini Tablets in Chocolate Pudding; Analysis was performed for etrasimod 2 mg mini tablets in chocolate pudding vs etrasimod 2 mg clinical IR tablet using mixed effect model with sequence, period and treatment as fixed effects and participant within the sequence as a random effect; Test type: Equivalence — For bioequivalence, the 90% CIs of the adjusted geometric mean ratio of AUClast for etrasimod 2 mg mini tablets mixed with chocolate pudding (tests) compared with etrasimod 2 mg clinical IR tablet (reference) were required to be within the 80 to 125% range; Ratio of adjusted geometric means = 94.96, 90% CI 2-sided [91.69 to 98.34] — The ratio and 90% CIs are expressed as percentages
Statistical Analysis 3: Comparison: Etrasimod 2 mg IR Tablet vs Etrasimod 2 mg Mini Tablets in Water; Analysis was performed for etrasimod 2 mg mini tablets in water vs etrasimod 2 mg clinical IR tablet using mixed effect model with sequence, period and treatment as fixed effects and participant within the sequence as a random effect; Test type: Equivalence — For bioequivalence, the 90% CIs of the adjusted geometric mean ratio of AUClast for etrasimod 2 mg mini tablets mixed with water (tests) compared with etrasimod 2 mg clinical IR tablet (reference) were required to be within the 80 to 125% range; Ratio of adjusted geometric means = 85.86, 90% CI 2-sided [82.90 to 88.92] — The ratio and 90% CIs are expressed as percentages
Statistical Analysis 4: Comparison: Etrasimod 2 mg IR Tablet vs Etrasimod 2 mg Mini Tablets in Yogurt; Analysis was performed for etrasimod 2 mg mini tablets in yogurt vs etrasimod 2 mg clinical IR tablet using mixed effect model with sequence, period and treatment as fixed effects and participant within the sequence as a random effect; Test type: Equivalence — For bioequivalence, the 90% CIs of the adjusted geometric mean ratio of AUClast for etrasimod 2 mg mini tablets mixed with yogurt (tests) compared with etrasimod 2 mg clinical IR tablet (reference) were required to be within the 80 to 125% range; Ratio of adjusted geometric means = 93.24, 90% CI 2-sided [89.76 to 96.84] — The ratio and 90% CIs are expressed as percentages

2. Primary Outcome: Area Under the Concentration-time Curve From Time Zero Extrapolated to Infinity (AUCinf) of Etrasimod
Description: AUCinf was calculated as AUClast + (Clast*/kel), where Clast is the predicted plasma concentration at the last quantifiable time point from the log-linear regression analysis, and kel is the terminal phase rate constant calculated by a linear regression of the loglinear concentration-time curve.
Time Frame: At pre-dose and 1, 2, 4, 6, 8, 12, 24, 48, 72, 96, 120, 144, and 168 hours post-dose on Day 1 of each period
Population: PK parameter analysis set included all participants who took at least 1 dose of study intervention and in whom at least 1 of the PK parameters of interest were reported.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*hr/mL
Arm/Group | Etrasimod 2 mg IR Tablet | Etrasimod 2 mg Mini Tablets in Applesauce | Etrasimod 2 mg Mini Tablets in Chocolate Pudding | Etrasimod 2 mg Mini Tablets in Water | Etrasimod 2 mg Mini Tablets in Yogurt
Number analyzed (Participants) | 16 | 15 | 16 | 16 | 16
ng*hr/mL | 1694 (26) | 1594 (20) | 1605 (19) | 1447 (23) | 1580 (22)
Statistical Analysis 1: Comparison: Etrasimod 2 mg IR Tablet vs Etrasimod 2 mg Mini Tablets in Applesauce; Analysis was performed for etrasimod 2 mg mini tablets in applesauce vs etrasimod 2 mg clinical IR tablet using mixed effect model with sequence, period and treatment as fixed effects and participant within the sequence as a random effect; Test type: Equivalence — For bioequivalence, the 90% CIs of the adjusted geometric mean ratio of AUCinf for etrasimod 2 mg mini tablets mixed with applesauce (tests) compared with etrasimod 2 mg clinical IR tablet (reference) were required to be within the 80 to 125% range; Ratio of adjusted geometric means = 94.36, 90% CI 2-sided [90.97 to 97.89] — The ratio and 90% CIs are expressed as percentages
Statistical Analysis 2: Comparison: Etrasimod 2 mg IR Tablet vs Etrasimod 2 mg Mini Tablets in Chocolate Pudding; [analysis description as in outcome 1, analysis 2]; Test type: Equivalence — For bioequivalence, the 90% CIs of the adjusted geometric mean ratio of AUCinf for etrasimod 2 mg mini tablets mixed with chocolate pudding (tests) compared with etrasimod 2 mg clinical IR tablet (reference) were required to be within the 80 to 125% range; Ratio of adjusted geometric means = 94.75, 90% CI 2-sided [91.41 to 98.20] — The ratio and 90% CIs are expressed as percentages
Statistical Analysis 3: Comparison: Etrasimod 2 mg IR Tablet vs Etrasimod 2 mg Mini Tablets in Water; [analysis description as in outcome 1, analysis 3]; Test type: Equivalence — For bioequivalence, the 90% CIs of the adjusted geometric mean ratio of AUCinf for etrasimod 2 mg mini tablets mixed with water (tests) compared with etrasimod 2 mg clinical IR tablet (reference) were required to be within the 80 to 125% range; Ratio of adjusted geometric means = 85.44, 90% CI 2-sided [82.43 to 88.55] — The ratio and 90% CIs are expressed as percentages
Statistical Analysis 4: Comparison: Etrasimod 2 mg IR Tablet vs Etrasimod 2 mg Mini Tablets in Yogurt; [analysis description as in outcome 1, analysis 4]; Test type: Equivalence — For bioequivalence, the 90% CIs of the adjusted geometric mean ratio of AUCinf for etrasimod 2 mg mini tablets mixed with yogurt (tests) compared with etrasimod 2 mg clinical IR tablet (reference) were required to be within the 80 to 125% range; Ratio of adjusted geometric means = 93.28, 90% CI 2-sided [89.61 to 97.10] — The ratio and 90% CIs are expressed as percentages

3. Primary Outcome: Maximum Observed Plasma Concentration (Cmax) for Etrasimod
Time Frame: At pre-dose and 1, 2, 4, 6, 8, 12, 24, 48, 72, 96, 120, 144, and 168 hours post-dose on Day 1 of each period
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Nanogram per milliliter
Arm/Group | Etrasimod 2 mg IR Tablet | Etrasimod 2 mg Mini Tablets in Applesauce | Etrasimod 2 mg Mini Tablets in Chocolate Pudding | Etrasimod 2 mg Mini Tablets in Water | Etrasimod 2 mg Mini Tablets in Yogurt
Number analyzed (Participants) | 16 | 15 | 16 | 16 | 16
Nanogram per milliliter | 43.18 (22) | 40.44 (19) | 40.03 (18) | 37.67 (18) | 39.98 (21)
Statistical Analysis 1: Comparison: Etrasimod 2 mg IR Tablet vs Etrasimod 2 mg Mini Tablets in Applesauce; [analysis description as in outcome 2, analysis 1]; Test type: Equivalence — For bioequivalence, the 90% CIs of the adjusted geometric mean ratio of Cmax for etrasimod 2 mg mini tablets mixed with applesauce (tests) compared with etrasimod 2 mg clinical IR tablet (reference) were required to be within the 80 to 125% range; Ratio of adjusted geometric means = 94.70, 90% CI 2-sided [90.38 to 99.22] — The ratio and 90% CIs are expressed as percentages
Statistical Analysis 2: Comparison: Etrasimod 2 mg IR Tablet vs Etrasimod 2 mg Mini Tablets in Chocolate Pudding; [analysis description as in outcome 1, analysis 2]; Test type: Equivalence — For bioequivalence, the 90% CIs of the adjusted geometric mean ratio of Cmax for etrasimod 2 mg mini tablets mixed with chocolate pudding (tests) compared with etrasimod 2 mg clinical IR tablet (reference) were required to be within the 80 to 125% range; Ratio of adjusted geometric means = 92.72, 90% CI 2-sided [88.59 to 97.04] — The ratio and 90% CIs are expressed as percentages
Statistical Analysis 3: Comparison: Etrasimod 2 mg IR Tablet vs Etrasimod 2 mg Mini Tablets in Water; [analysis description as in outcome 1, analysis 3]; Test type: Equivalence — For bioequivalence, the 90% CIs of the adjusted geometric mean ratio of Cmax for etrasimod 2 mg mini tablets mixed with water (tests) compared with etrasimod 2 mg clinical IR tablet (reference) were required to be within the 80 to 125% range; Ratio of adjusted geometric means = 87.24, 90% CI 2-sided [83.35 to 91.31] — The ratio and 90% CIs are expressed as percentages
Statistical Analysis 4: Comparison: Etrasimod 2 mg IR Tablet vs Etrasimod 2 mg Mini Tablets in Yogurt; [analysis description as in outcome 1, analysis 4]; Test type: Equivalence — For bioequivalence, the 90% CIs of the adjusted geometric mean ratio of Cmax for etrasimod 2 mg mini tablets mixed with yogurt (tests) compared with etrasimod 2 mg clinical IR tablet (reference) were required to be within the 80 to 125% range; Ratio of adjusted geometric means = 92.59, 90% CI 2-sided [88.24 to 97.17] — The ratio and 90% CIs are expressed as percentages

4. Secondary Outcome: Change From Baseline in Heart Rate at 1, 2, 3, 4, 5, 6, 8 and 24 Hours on Day 1
Description: Heart rate was measured in beats per minute.
Time Frame: Baseline, 1, 2, 3, 4, 5, 6, 8 and 24 hours post dose on Day 1
Population: SAS included all participants who took at least 1 dose of study intervention. Participants were analyzed according to the product they actually received.
Measure: Mean (Standard Deviation); unit: Beats per minute
Arm/Group | Etrasimod 2 mg IR Tablet | Etrasimod 2 mg Mini Tablets in Applesauce | Etrasimod 2 mg Mini Tablets in Chocolate Pudding | Etrasimod 2 mg Mini Tablets in Water | Etrasimod 2 mg Mini Tablets in Yogurt
Number analyzed (Participants) | 16 | 15 | 16 | 16 | 16
Beats per minute
  At 1 hour | -6.3 (4.08) | -6.0 (3.85) | -6.9 (7.12) | -3.9 (3.75) | -5.1 (4.32)
  At 2 hours | -10.4 (3.03) | -9.6 (2.38) | -11.5 (6.55) | -9.8 (4.51) | -10.5 (4.62)
  At 3 hours | -10.8 (4.60) | -9.9 (2.97) | -12.1 (7.41) | -10.1 (5.07) | -10.3 (4.39)
  At 4 hours | -9.9 (4.84) | -8.8 (3.21) | -11.0 (7.08) | -8.7 (4.32) | -11.0 (3.85)
  At 5 hours | -4.1 (4.52) | -2.5 (3.27) | -5.1 (6.98) | -2.3 (4.27) | -4.4 (4.46)
  At 6 hours | -3.4 (4.67) | -2.0 (3.96) | -4.4 (6.33) | -3.1 (3.61) | -2.6 (3.88)
  At 8 hours | -5.3 (4.75) | -4.3 (3.63) | -5.9 (6.48) | -4.9 (6.10) | -3.8 (7.99)
  At 24 hours | -6.4 (3.14) | -5.6 (6.19) | -7.4 (7.38) | -6.8 (4.62) | -6.8 (5.80)

5. Secondary Outcome: Number of Participants With Treatment Emergent Adverse Events (TEAEs)
Description: An adverse event (AE) was any untoward medical occurrence in a participant or clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. TEAEs were any AEs that occurred following start of treatment. A serious adverse event (SAE) was defined as any untoward medical occurrence that at any dose, met one or more of the criteria: resulted in death, life-threatening, required inpatient hospitalization or prolongation of existing hospitalization, results in persistent or significant disability/incapacity, congenital anomaly/birth defect. AEs included SAEs and all non-SAEs.
Time Frame: From start of study treatment up to 28-35 days after last dose of study treatment (maximum up to 72 days)
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | Etrasimod 2 mg IR Tablet | Etrasimod 2 mg Mini Tablets in Applesauce | Etrasimod 2 mg Mini Tablets in Chocolate Pudding | Etrasimod 2 mg Mini Tablets in Water | Etrasimod 2 mg Mini Tablets in Yogurt
Number analyzed (Participants) | 16 | 15 | 16 | 16 | 16
Participants | 7 | 10 | 9 | 8 | 11

6. Secondary Outcome: Number of Participants With Clinical Laboratory Abnormalities
Description: Clinical laboratory abnormalities test criteria included haematology: lymphocytes (10^3/ mm^3) and lymphocytes/leukocytes percentage (%) less than (<) 0.8* lower limit of normal (LLN), neutrophils, eosinophils, monocytes (10^3/mm^3), eosinophils/leukocytes monocytes/leukocytes (%) more than (>) 1.2* upper limit of normal (ULN); clinical chemistry: bicarbonate milliequivalents per liter (mEq/L) > 1.1* ULN; Urinalysis: urine hemoglobin, nitrite, leukocyte esterase greater than or equal to (>=) 1 and squamous epithelial cells /low power field (/LPF) > 4. Number of participants meeting any clinical laboratory abnormalities criteria is reported in this outcome measure.
Time Frame: Up to Day 45
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | Etrasimod 2 mg IR Tablet | Etrasimod 2 mg Mini Tablets in Applesauce | Etrasimod 2 mg Mini Tablets in Chocolate Pudding | Etrasimod 2 mg Mini Tablets in Water | Etrasimod 2 mg Mini Tablets in Yogurt
Number analyzed (Participants) | 16 | 15 | 16 | 16 | 16
Participants | 5 | 10 | 8 | 5 | 6

7. Secondary Outcome: Number of Participants According to Categorization of Vital Signs Results
Description: Supine blood pressure (SBP) and pulse rate (PR) were measured. Vital sign criteria included: Systolic BP: <90 millimeter of mercury [mmHg]; Systolic BP change from baseline: maximum increase and decrease >=30 mmHg; Diastolic BP < 50 mmHg; Diastolic BP change from baseline: maximum decrease and increase >=20 mmHg; pulse rate <40 and >120 beats per minute.
Time Frame: Up to Day 45
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | Etrasimod 2 mg IR Tablet | Etrasimod 2 mg Mini Tablets in Applesauce | Etrasimod 2 mg Mini Tablets in Chocolate Pudding | Etrasimod 2 mg Mini Tablets in Water | Etrasimod 2 mg Mini Tablets in Yogurt
Number analyzed (Participants) | 16 | 15 | 16 | 16 | 16
Participants
  Supine Systolic Blood Pressure (mmHg) Value <90 | 0 | 2 | 1 | 1 | 1
  Supine Systolic Blood Pressure (mmHg) Value Change >= 30 Increase | 0 | 0 | 0 | 1 | 0
  Supine Systolic Blood Pressure (mmHg) Value Change >= 30 decrease | 0 | 0 | 0 | 0 | 0
  Supine Diastolic Blood Pressure (mmHg) Value <50 | 0 | 0 | 0 | 0 | 0
  Supine Diastolic Blood Pressure (mmHg) Value >= 20 increase | 0 | 0 | 0 | 1 | 0
  Supine Diastolic Blood Pressure (mmHg) Value >= 20 decrease | 0 | 0 | 3 | 0 | 0
  Supine Pulse Rate (beats/min) Value <40 | 0 | 1 | 0 | 0 | 0
  Supine Pulse Rate (beats/min) Value >120 | 0 | 0 | 0 | 0 | 0

8. Secondary Outcome: Number of Participants According to Categorization of Electrocardiograms (ECGs) Findings
Description: Standard 12-lead ECGs were used to measure PR interval, QT interval, QTc corrected using Fridericia's formula (QTcF), and QRS complex. ECG abnormalities were categorized as: QTcF interval, aggregate (milliseconds [msec]) 450 < Value <= 480, 480 < value <= 500, value > 500; 30 <= Change <= 60; Change > 60. Participants with any ECG abnormality criteria were reported in this outcome measure.
Time Frame: Up to Day 45
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | Etrasimod 2 mg IR Tablet | Etrasimod 2 mg Mini Tablets in Applesauce | Etrasimod 2 mg Mini Tablets in Chocolate Pudding | Etrasimod 2 mg Mini Tablets in Water | Etrasimod 2 mg Mini Tablets in Yogurt
Number analyzed (Participants) | 16 | 15 | 16 | 16 | 16
Participants
  QTcF interval aggregate (Msec): 450 < Value <= 480 | 0 | 0 | 0 | 0 | 0
  QTcF interval aggregate (Msec): 480 < Value <= 500 | 0 | 0 | 0 | 0 | 0
  QTcF interval aggregate (Msec): Value > 500 | 0 | 0 | 0 | 0 | 0
  QTcF interval aggregate (Msec): 30 <= Change <= 60 | 1 | 0 | 0 | 0 | 0
  QTcF interval aggregate (Msec): Change > 60 | 0 | 0 | 0 | 0 | 0

9. Secondary Outcome: Assessment of Mouth Feel Based on Palatability Questionnaire
Description: Participants were required to answer mouth feel (such as grittiness, stickiness, waxiness) of the product tasted. The score ranged from 0 (favorable) to 100 (not favorable), where higher scores indicated worse mouth feel.
Time Frame: At 1, 5, 10 and 20 minutes after tasting dose in each vehicle on Day 1 of each period
Population: SAS included all participants who took at least 1 dose of study intervention. Participants were analyzed according to the product they actually received. As specified in protocol, data for 2mg-IR tablet (Reference) arm was not evaluated because it was planned to assess palatability of mini tabs in each vehicle (applesauce, chocolate pudding, water and yogurt) [Test]. Here "Number Analyzed" refers to the number of participants evaluable for the specified rows.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Etrasimod 2 mg Mini Tablets in Applesauce | Etrasimod 2 mg Mini Tablets in Chocolate Pudding | Etrasimod 2 mg Mini Tablets in Water | Etrasimod 2 mg Mini Tablets in Yogurt
Number analyzed (Participants) | 15 | 16 | 16 | 16
Score on a scale
  At 1 minute | 8.0 (10.34) | 5.0 (7.21) | 9.6 (17.14) | 9.3 (10.03)
  At 5 minutes | 6.9 (9.93) | 4.7 (5.36) | 8.1 (15.84) | 8.4 (12.46)
  At 10 minutes: number analyzed (Participants) | 15 | 14 | 13 | 16
  At 10 minutes | 5.6 (10.27) | 6.6 (7.12) | 8.9 (18.04) | 7.4 (9.16)
  At 20 minutes | 7.0 (14.59) | 5.6 (5.23) | 8.8 (16.22) | 4.8 (6.61)

10. Secondary Outcome: Assessment of Bitterness Based on Palatability Questionnaire
Description: Participants were required to tell about the degree of bitterness of the product tasted. The score ranged from 0 (favorable) to 100 (not favorable), where higher scores indicated worse bitterness.
Time Frame: At 1, 5, 10 and 20 minutes after tasting dose in each vehicle on Day 1 of each period
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Etrasimod 2 mg Mini Tablets in Applesauce | Etrasimod 2 mg Mini Tablets in Chocolate Pudding | Etrasimod 2 mg Mini Tablets in Water | Etrasimod 2 mg Mini Tablets in Yogurt
Number analyzed (Participants) | 15 | 16 | 16 | 16
Score on a scale
  At 1 minute | 12.3 (17.26) | 4.3 (5.69) | 9.4 (17.02) | 8.9 (15.09)
  At 5 minutes | 5.0 (7.41) | 4.1 (4.92) | 8.3 (16.07) | 7.9 (12.39)
  At 10 minutes: number analyzed (Participants) | 15 | 14 | 13 | 16
  At 10 minutes | 4.2 (4.86) | 5.5 (6.53) | 9.9 (18.52) | 7.8 (11.49)
  At 20 minutes | 3.5 (3.91) | 4.2 (4.65) | 9.3 (17.50) | 4.3 (5.49)

11. Secondary Outcome: Assessment of Tongue/Mouth Burns Based on Palatability Questionnaire
Description: Participants were required to tell about the degree of palatability attribute of tongue/mouth burns of the product tasted. The score ranged from 0 (favorable) to 100 (not favorable), where higher scores indicated more tongue/mouth burns.
Time Frame: At 1, 5, 10 and 20 minutes after tasting dose in each vehicle on Day 1 of each period
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Etrasimod 2 mg Mini Tablets in Applesauce | Etrasimod 2 mg Mini Tablets in Chocolate Pudding | Etrasimod 2 mg Mini Tablets in Water | Etrasimod 2 mg Mini Tablets in Yogurt
Number analyzed (Participants) | 15 | 16 | 16 | 16
Score on a scale
  At 1 minute | 3.4 (3.81) | 2.7 (3.48) | 3.9 (4.04) | 4.8 (5.26)
  At 5 minutes | 3.1 (3.76) | 3.1 (3.26) | 3.8 (3.34) | 3.4 (4.26)
  At 10 minutes: number analyzed (Participants) | 15 | 14 | 13 | 16
  At 10 minutes | 3.0 (3.80) | 3.6 (3.44) | 4.2 (3.36) | 3.6 (4.10)
  At 20 minutes | 3.1 (3.56) | 4.3 (4.44) | 7.1 (10.16) | 3.0 (2.63)

12. Secondary Outcome: Assessment of Likeness of Throat Burn Based on Palatability Questionnaire
Description: Participants were required to tell the palatability attribute of throat burn of the product tasted. The score ranged from 0 (favorable) to 100 (not favorable), where higher scores indicated more throat burn.
Time Frame: At 1, 5, 10 and 20 minutes after tasting dose in each vehicle on Day 1 of each period
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Etrasimod 2 mg Mini Tablets in Applesauce | Etrasimod 2 mg Mini Tablets in Chocolate Pudding | Etrasimod 2 mg Mini Tablets in Water | Etrasimod 2 mg Mini Tablets in Yogurt
Number analyzed (Participants) | 15 | 16 | 16 | 16
Score on a scale
  At 1 minute | 6.9 (13.48) | 3.4 (3.77) | 4.0 (4.35) | 5.3 (7.04)
  At 5 minutes | 6.6 (12.16) | 3.6 (3.67) | 3.7 (3.46) | 6.8 (12.03)
  At 10 minutes: number analyzed (Participants) | 15 | 14 | 13 | 16
  At 10 minutes | 6.3 (12.12) | 5.3 (7.04) | 10.2 (18.69) | 8.1 (17.98)
  At 20 minutes | 6.2 (12.32) | 3.6 (3.95) | 13.6 (25.19) | 8.8 (17.28)

13. Secondary Outcome: Assessment of Overall Liking Based on Palatability Questionnaire
Description: Participants were required to tell the palatability attribute of overall liking of the product tasted. The score ranged from 0 (favorable) to 100 (not favorable), where higher scores indicated less overall liking.
Time Frame: At 1, 5, 10 and 20 minutes after tasting dose in each vehicle on Day 1 of each period
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Etrasimod 2 mg Mini Tablets in Applesauce | Etrasimod 2 mg Mini Tablets in Chocolate Pudding | Etrasimod 2 mg Mini Tablets in Water | Etrasimod 2 mg Mini Tablets in Yogurt
Number analyzed (Participants) | 15 | 16 | 16 | 16
Score on a scale
  At 1 minute | 8.9 (13.58) | 3.8 (4.90) | 8.1 (16.69) | 10.4 (14.24)
  At 5 minutes | 6.8 (12.20) | 4.4 (3.76) | 7.9 (16.55) | 10.1 (16.62)
  At 10 minutes: number analyzed (Participants) | 15 | 14 | 13 | 16
  At 10 minutes | 6.5 (12.25) | 5.4 (4.78) | 9.2 (19.10) | 10.1 (18.64)
  At 20 minutes | 6.6 (12.55) | 4.3 (4.01) | 9.2 (17.70) | 9.8 (16.31)

ADVERSE EVENTS:
Time Frame: From start of study treatment up to 28-35 days after last dose of study treatment (maximum up to 72 days)
Arm/Group | Etrasimod 2 mg IR Tablet | Etrasimod 2 mg Mini Tablets in Applesauce | Etrasimod 2 mg Mini Tablets in Chocolate Pudding | Etrasimod 2 mg Mini Tablets in Water | Etrasimod 2 mg Mini Tablets in Yogurt
All-Cause Mortality (participants affected / at risk) | 0/16 | 0/15 | 0/16 | 0/16 | 0/16
Serious Adverse Events (participants affected / at risk) | 0/16 | 0/15 | 0/16 | 0/16 | 0/16
Other Adverse Events (participants affected / at risk) | 7/16 | 10/15 | 9/16 | 8/16 | 11/16
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Etrasimod 2 mg IR Tablet (N=16) | Etrasimod 2 mg Mini Tablets in Applesauce (N=15) | Etrasimod 2 mg Mini Tablets in Chocolate Pudding (N=16) | Etrasimod 2 mg Mini Tablets in Water (N=16) | Etrasimod 2 mg Mini Tablets in Yogurt (N=16)
Atrioventricular block first degree (Cardiac disorders) | 1 | 0 | 1 | 1 | 1
Ear pain (Ear and labyrinth disorders) | 0 | 0 | 1 | 0 | 0
Asthenopia (Eye disorders) | 0 | 1 | 0 | 0 | 0
Ocular hyperaemia (Eye disorders) | 0 | 1 | 1 | 0 | 0
Photopsia (Eye disorders) | 0 | 0 | 0 | 1 | 0
Vision blurred (Eye disorders) | 1 | 1 | 0 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Change of bowel habit (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Constipation (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Dyspepsia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 2
Glossodynia (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
Lip dry (Gastrointestinal disorders) | 2 | 0 | 1 | 1 | 2
Nausea (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Tongue ulceration (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Toothache (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Asthenia (General disorders) | 0 | 0 | 0 | 0 | 1
Fatigue (General disorders) | 1 | 1 | 2 | 2 | 3
Influenza like illness (General disorders) | 0 | 0 | 1 | 0 | 0
Puncture site erythema (General disorders) | 2 | 0 | 0 | 0 | 0
Vessel puncture site erythema (General disorders) | 0 | 0 | 0 | 1 | 0
Vessel puncture site haematoma (General disorders) | 3 | 0 | 2 | 1 | 0
Influenza (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Nasopharyngitis (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Oral herpes (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Post procedural haematoma (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0
Skin laceration (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0
Sunburn (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0
Burning sensation (Nervous system disorders) | 0 | 0 | 1 | 0 | 0
Dizziness (Nervous system disorders) | 0 | 1 | 1 | 0 | 4
Dizziness postural (Nervous system disorders) | 0 | 0 | 0 | 1 | 0
Dysgeusia (Nervous system disorders) | 1 | 0 | 0 | 0 | 0
Headache (Nervous system disorders) | 1 | 2 | 0 | 0 | 2
Presyncope (Nervous system disorders) | 0 | 0 | 0 | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0
Oropharyngeal discomfort (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0 | 0 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1
Acne (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0
Dermal cyst (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 2 | 0 | 0 | 0
Erythema (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 2
Rash macular (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0
Rosacea (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0
Skin exfoliation (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0
Haematoma (Vascular disorders) | 1 | 0 | 0 | 0 | 0
Hot flush (Vascular disorders) | 0 | 0 | 0 | 0 | 1

LIMITATIONS AND CAVEATS:
Any untoward findings identified on physical examination during the active collection period were captured as adverse events, if those findings met the definition of an AE.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publication until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.

DOCUMENTS (2):
  • Study Protocol (2023-06-01): https://cdn.clinicaltrials.gov/large-docs/02/NCT05956002/Prot_000.pdf
  • Statistical Analysis Plan (2023-05-25): https://cdn.clinicaltrials.gov/large-docs/02/NCT05956002/SAP_001.pdf